CLINICAL TRIAL: NCT01557452
Title: An Open-Label Extension of the Dose Finding Study (DSC/08/2357/36) in Patients With Polyarticular Course Juvenile Idiopathic Arthritis (Poly JIA)
Brief Title: Open-Label Extension of the Dose Finding Study (DSC/08/2357/36) in Patients With Poly Juvenile Idiopathic Arthritis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Previous study DSC/08/2357/36 did not show efficacy for Givinostat in JIA. Sponsor decision to stop development of Givinostat in polyarticular course Juvenile Idiopathic Arthritis wasn't related to any tolerability concerns.
Sponsor: Italfarmaco (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSC/11/2357/42; 2011-003341-18 (EudraCT Number)
Record Dates: First submitted 2012-03-14; First posted 2012-03-19 (Estimated); Results first posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-03

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: JIA
MeSH Terms: conditions — Arthritis, Juvenile | interventions — givinostat; givinostat hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Givinostat (Experimental): Patient received the dose of 0.75 mg/kg BID from December 28th, 2011 to January 27th, 2014
  Interventions: Drug: Givinostat

INTERVENTIONS:
Drug: Givinostat — ready-to-use oral suspension, administered in fed condition and on a outpatient basis, especially intended for paediatric patients
  Other Names: ITF2357

SUMMARY:
Primary Objective of the study:

the purpose of this extension study was to determine the safety of Givinostat in a long term treatment of patients who participated in DSC/08/2357/36 study with good results (clinical benefit at least pediACR30 response);

DETAILED DESCRIPTION:
Givinostat is expected to exert a clinically relevant therapeutic effect on polyarticular JIA through the inhibition of the production/release of pro-inflammatory cytokines, such as IL-1β, IL-6 and TNFα, which are involved in the pathogenesis of the arthritic process.

ELIGIBILITY:
Inclusion Criteria:

* subjects who had successfully completed the previous Dose Finding Study and were fully compliant to the inclusion/exclusion criteria described in the previous DSC/08/2357/36

Exclusion Criteria:

* patients with fever related to JIA or other systemic features of JIA during 12 months before entering the study
* active bacterial or mycotic infection requiring antimicrobial treatment
* episode of macrophage activation syndrome over the last 6 months
* baseline prolongation of QT/QTc interval, use of concomitant medications that prolong the QT/QTc interval or history of additional risk factors for TdP.
* clinically significant cardiovascular disease
* clinically significant illness i.e. any condition that in the opinion of the Investigator places the patient to unacceptable risk for adverse outcome if he/she were to participate in the study
* psychiatric illness/social situation that would limit compliance with study medication and protocol requirements
* inherited metabolic diseases
* presence of malignancy
* pregnancy or lactation
* positive blood test for HIV
* active EBV infection, active B and/or C hepatitis
* platelet count <100x10(9)/L

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2011-12-28 (Actual); Primary Completion 2014-01-27 (Actual); Study Completion 2014-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pavla Dolezalova, MD, Principal Investigator — General Faculty Hospital Department of Pediatrics and Adolescent Medicine, Praha, Czech Republic
Locations (1):
- 1st Faculty of Medicine and General Faculty Hospital, Prague, Czechia

RESULTS

PARTICIPANT FLOW:
Groups:
- Givinostat: Givinostat: oral suspension, 0,75 mg/Kg b.i.d. in fed conditions
Period: Overall Study
Arm/Group | Givinostat
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Givinostat
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Czechia | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAE) and Adverse Events (AE) of Interest
Description: During the entire study period it was reported only one adverse event considered not drug related by the investigator (Mild flu at week 107 of study treatment).
  No action was taken and the patient recovered spontaneously
Time Frame: Through end of treatment, up to 108 weeks.
Measure: Number; unit: participants
Arm/Group | Givinostat
Number analyzed (Participants) | 1
participants
  non serious AE | 1
  serious AE | 0

2. Secondary Outcome: Number of Patients Who Maintained PedACR30 Response
Description: This is an open-label treatment extension of the 2010-019094-15 study, an antecedent dose-ranging trial of Givinostat ready-to-use oral suspension formulation. Eligible patients were those who had completed the previous study achieving a clinical benefit, i.e. patients achieving at least an ACR Paediatric 30 (PedACR30).
  PedACR30 is defined as at least a 30% improvement from baseline in any three of the following six variables in juvenile idiopathic arthritis (JIA) patients, with no more than one variable worsening by more than 30%:
  * physician's global assessment of disease activity;
  * parent/guardian's or patient's global assessment of overall wellbeing;
  * functional ability;
  * number of joints with active arthritis;
  * number of joints with limited range of motion;
  * ESR.
  (ACR stands for American College of Rheumatology)
Time Frame: At weeks 48, 60 and 108
Measure: Number; unit: participants
Arm/Group | Givinostat
Number analyzed (Participants) | 1
participants
  week 48 | 1
  week 60 | 0
  week 108 | 1

3. Secondary Outcome: Number of Patients Who Reached PedACR70 Response
Description: This is an open-label treatment extension of the 2010-019094-15 study, an antecedent dose-ranging trial of Givinostat ready-to-use oral suspension formulation. Eligible patients were those who had completed the previous study achieving a clinical benefit, i.e. patients achieving at least an ACR Paediatric 30 (PedACR30).
  PedACR70 is defined as at least a 70% improvement from baseline in any three of the following six variables in juvenile idiopathic arthritis (JIA) patients, with no more than one variable worsening by more than 30%:
  * physician's global assessment of disease activity;
  * parent/guardian's or patient's global assessment of overall wellbeing;
  * functional ability;
  * number of joints with active arthritis;
  * number of joints with limited range of motion;
  * ESR.
  (ACR stands for American College of Rheumatology)
Time Frame: At weeks 48, 60 and 108
Measure: Number; unit: participants
Arm/Group | Givinostat
Number analyzed (Participants) | 1
participants
  week 48 | 0
  week 60 | 1
  week 108 | 0

ADVERSE EVENTS:
Time Frame: Through end of treatment, up to 108 weeks.
Arm/Group | Givinostat
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Givinostat (N=1)
Influenza (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No